CLINICAL TRIAL: NCT03768180
Title: INfecTive ENdocarditis After Transcatheter Aortic Valve Replacement (TAVR) a National SwEdish Study (INTENSE)
Brief Title: Infective Endocarditis After TAVR
Acronym: INTENSE
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: IETAVR
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2019-03

CONDITIONS: Infective Endocarditis of Aortic Valve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with infective endocarditis: All patients diagnosed with infective endocarditis after TAVR

SUMMARY:
This study aims at studying the frequency of infective endocarditis after transcatheter aortic valve replacement/implantation

DETAILED DESCRIPTION:
Since the start of transcatheter aortic valve implnatations/replacements (TAVR/TAVI) implantations in Sweden in 2008 all procedures have been added to a national database, which now contains 4500+ procedures. At the same time, all admissions to the hospital is also recorded with diagnosis in a separate database. We intend to make a nation-wide complete follow up of all TAVR/TAVI patients in swede that has received the diagnosis of infective endocarditis after the implantation. In addition data will also be collected from the national endocarditis database for detailed information of the cases.

ELIGIBILITY:
Inclusion Criteria:

All patients that has under TAVR/TAVI in Sweden between 2008 and 2018

Exclusion Criteria:

Patients unable to follow up due to emigration or missing social security number

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that has under TAVR/TAVI in Sweden between 2008 and 2018
Sampling Method: Probability Sample
Enrollment: 4600 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Infective Endocarditis | 5 year
  Patients that have suffered an infective endocarditis will be described, where survival is one important variable

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjursten H, Rasmussen M, Nozohoor S, Gotberg M, Olaison L, Ruck A, Ragnarsson S. Infective endocarditis after transcatheter aortic valve implantation: a nationwide study. Eur Heart J. 2019 Oct 14;40(39):3263-3269. doi: 10.1093/eurheartj/ehz588. PMID 31433472